CLINICAL TRIAL: NCT00882765
Title: A Pre-Surgical, Randomized Clinical Trial of Genistein in Resectable Pancreatic Adenocarcinoma
Brief Title: Genistein in Treating Patients With Pancreatic Cancer That Can Be Removed by Surgery
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study has been closed due to no accrual.
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000639616; UCLA-0808100; NCI-2010-00242 (Registry Identifier: CTRP)
Record Dates: First submitted 2009-04-15; First posted 2009-04-16 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2012-07

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; stage I pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Genistein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive neoadjuvant oral genistein once daily for 2 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Dietary Supplement: genistein
- No intervention (No Intervention): Patients receive no specific neoadjuvant therapy.

INTERVENTIONS:
Dietary Supplement: genistein — Given orally
  Arms: Arm I

SUMMARY:
RATIONALE: Genistein may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving genistein before surgery may be an effective treatment for pancreatic cancer.

PURPOSE: This randomized phase II trial is studying genistein to see how well it works in treating patients with pancreatic cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine changes in microvessel density of the tumor specimen after 2 weeks of treatment with genistein in patients with resectable pancreatic adenocarcinoma.

Secondary

* To evaluate the safety and tolerability of genistein in these patients by looking at the impact of genistein on pancreatic cancer angiogenesis and on the angiogenic factors VEGF, CXCL1, CXCL5, and CXCL8.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive neoadjuvant oral genistein once daily for 2 weeks in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive no specific neoadjuvant therapy. In both arms, patients undergo surgical resection in week 3.

Blood, urine, and tissue samples are collected at baseline and at the time of surgery for laboratory biomarker studies. Samples are analyzed for VEGF, CXCL1, CXCL5, and CXCL8 by ELISA and for genistein by mass spectrometry.

ELIGIBILITY:
Inclusion Criteria:

* Adults over the age of 18 capable of giving informed consent
* resectable pancreatic mass, known or presumed to be primary pancreatic adenocarcinoma. Patients whose initial biopsy do not show adenocarcinoma will not receive the study drug.
* ECOG preformance status 0-2.
* Negative pregnancy test prior to initiation of treatment and adequate contraception throughout treatment.

Exclusion criteria:

* comorbid disease or medical condition that would impair the ability of the patient to receive or comply with the study protocol
* hypersensitivity to genistein or to any of the excipients of genistein
* prior chemotherapy or radiotherapy for pancreatic adenocarcinoma
* concomitant use of warfarin, tamoxifen, or raloxifene.
* pregnancy or inadequate contraception.
* lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-05; Primary Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Changes in microvessel density of tumor specimen after 2 weeks of treatment with genistein | 2 weeks

SECONDARY OUTCOMES:
To evaluate the impact of genistein on the angiogenic factors VEGF, CXCL1, CXCL5, and CXCL8 | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Edward Garon, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA, Los Angeles, California, United States